CLINICAL TRIAL: NCT00000699
Title: A Phase I/II Trial of Ribavirin (With Escalation) + Isoprinosine in Asymptomatic HIV-Viremic Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: NS 403
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-08-26 (Estimated); Status verified 2003-04

CONDITIONS: HIV Infections
Keywords: Ribavirin; Inosine Pranobex; Dose-Response Relationship, Drug; Drug Evaluation; Drug Therapy, Combination; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — Inosine Pranobex; Ribavirin

INTERVENTIONS:
Drug: Inosine pranobex
Drug: Ribavirin

SUMMARY:
To determine the safety and effectiveness of treatment with ribavirin (RBV) plus isoprinosine (INPX) in preventing the development of AIDS in patients infected with the AIDS virus (HIV). Also to determine the maximal dose of RBV that can be tolerated by HIV-infected patients when RBV is given with INPX. The patients may or may not have generalized lymphadenopathy syndrome (LAS). RBV has prevented the development of AIDS in some HIV-infected patients with LAS and INPX has stimulated the immune system of patients infected with HIV. The immune system fights infections in the human body, and the HIV attacks T cells that are an important part of the immune system. Reports from individual cases treated with both RBV and INPX suggest that clinical improvements occurred in HIV-infected patients, but there is no reliable information on the safety and effectiveness of this drug combination in such patients.

DETAILED DESCRIPTION:
RBV has prevented the development of AIDS in some HIV-infected patients with LAS and INPX has stimulated the immune system of patients infected with HIV. The immune system fights infections in the human body, and the HIV attacks T cells that are an important part of the immune system. Reports from individual cases treated with both RBV and INPX suggest that clinical improvements occurred in HIV-infected patients, but there is no reliable information on the safety and effectiveness of this drug combination in such patients.

All patients take INPX capsules 4 times a day and RBV capsules 2 or 3 times a day. The first group of patients take the dose of RBV shown to be effective in an earlier trial and subsequent groups take higher doses until toxic effects occur. The planned treatment period is 3 months, but further treatment may be allowed for patients showing improvement. Blood samples are taken from an arm vein and used to evaluate possible changes in the patient's immune system, any toxic effects that might be detected in the blood and possible changes in the presence of HIV in the blood.

ELIGIBILITY:
Inclusion Criteria

* It must be possible to culture HIV from peripheral blood lymphocytes on 2 consecutive screenings within 2 months of starting treatment.

Concurrent Medication:

Allowed:

* Systemic medications not listed in the Exclusion Concurrent Medications field considered necessary for the patient's medical management and which would not interfere with the study may be used, but such use must be documented.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Systemic steroids.
* Cytotoxic immunosuppressive medications.
* Any systemic experimental anti-HIV drug such as dideoxycytidine (ddC), foscarnet, ribavirin, isoprinosine, or zidovudine (AZT).
* Any other medication felt to be immunomodulatory or felt to exhibit significant hepatotoxicity or hematologic or renal toxicity by study investigators.

Prior Medication:

Excluded within 6 weeks of study entry:

* Systemic steroids.
* Cytotoxic immunosuppressive medications.
* Any systemic experimental anti-HIV drug such as dideoxycytidine (ddC), foscarnet, ribavirin, isoprinosine, or zidovudine (AZT).
* Any other medication felt to be immunomodulatory or felt to exhibit significant hepatotoxicity or hematologic or renal toxicity by study investigators.

Current active infections, known cardiac disease, or prior history of one of the following:

* Gout, uric acid urolithiasis, uric acid nephrolithiasis, or renal dysfunction.
* Neoplasms:
* Other than locally treated basal or squamous carcinoma.
* Cardiovascular:
* Myocardial infarction, cardiac arrhythmia, cardiomyopathy, or congestive heart failure.

Past or current history of CDC-defined AIDS including HIV encephalopathy and HIV wasting syndrome. Constitutional symptoms (CDC Group IV-A), neurologic symptoms (CDC Group IV-B), or any prior or current non-AIDS defining secondary infectious disease (CDC Group IV-C2). Grade 1 impairment on 2 or more items in the ACTG Micro Neuro-AIDS Assessment.

Active drug or alcohol abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20

CONTACTS AND LOCATIONS:
Overall Officials: Schulof RS, Study Chair
Locations (1):
- George Washington Univ Med Ctr, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Schulof R, Simon G, Parenti D, Sztein M, Meyer W, Paxton H. Phase I/II trial of ribavirin + isoprinosine in asymptomatic HIV viremic gay men. Int Conf AIDS. 1989 Jun 4-9;5:212 (abstract no ThBO2)
- [Background] Schulof RS, Parenti DM, Simon GL, Paxton H, Meyer WA 3rd, Schlesselman SB, Courtless J, LeLacheur S, Sztein MB. Clinical, virologic, and immunologic effects of combination therapy with ribavirin and isoprinosine in HIV-infected homosexual men. J Acquir Immune Defic Syndr (1988). 1990;3(5):485-92. PMID 1691287